CLINICAL TRIAL: NCT02691247
Title: A Prospective Randomized Placebo-Controlled Double Blind Clinical Trial to Evaluate the Safety and Efficacy of CLBS03 (Autologous Ex Vivo Expanded Polyclonal Regulatory T-cells) in Adolescents With Recent Onset Type 1 Diabetes Mellitus (T1DM)
Brief Title: Safety and Efficacy of CLBS03 in Adolescents With Recent Onset Type 1 Diabetes (The Sanford Project T-Rex Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Collaborators: Sanford Health (Other); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLBS03-P01
Record Dates: First submitted 2016-02-12; First posted 2016-02-25 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus
Keywords: T1DM; Type 1 Diabetes Mellitus; T regulatory cell; Immunotherapy; Cell therapy; T-Reg
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CLBS03 Low Dose (Experimental): A single infusion of CLBS03 Low Dose, a cell product comprised of autologous, ex vivo expanded regulatory T-cells resuspended in sterile USP (United States Pharmacopoeia) infusion solution.
  Interventions: Biological: CLBS03 Low Dose
- CLBS03 High Dose (Experimental): A single infusion of CLBS03 High Dose, a cell product comprised of autologous, ex vivo expanded regulatory T-cells resuspended in sterile USP infusion solution.
  Interventions: Biological: CLBS03 High Dose
- Placebo (Placebo Comparator): A single infusion of placebo, consisting of the infusion solution only
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CLBS03 Low Dose
  Arms: CLBS03 Low Dose
Biological: CLBS03 High Dose
  Arms: CLBS03 High Dose
Biological: Placebo
  Arms: Placebo

SUMMARY:
This clinical trial will explore the safety and effect of autologous ex vivo expanded polyclonal regulatory T-cells on beta cell function in patients, aged 8 to 17, with recent onset T1DM. Other measures of diabetes severity and the autoimmune response underlying T1DM will also be explored. Eligible subjects will receive a single infusion of CLBS03 (high or low dose) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged 8 to 17 years of age
* Diagnosis of T1DM within 100 days of receipt of study drug
* Positive for at least one islet cell autoantibody
* Peak MMTT-stimulated C-peptide level > 0.2 pmol/mL (at the screening visit)
* Weight of ≥30 kg
* Must agree to use a reliable and acceptable method of contraception for the duration of participation
* Willing and medically acceptable to postpone live vaccine immunizations for one year after infusion
* Written informed consent and written assent

Exclusion Criteria:

* Hemoglobin less than the lower limit of normal
* Leukocytes <3,000/μL; neutrophils <1,500/μL; lymphocytes <800/μL; platelets <100,000/μL
* Regulatory T-cells present in peripheral blood at <20 cells per μL
* Current or ongoing use of non-insulin pharmaceuticals (that may affect glycemic control)
* Current or anticipated use of systemic corticosteroids or other immunomodulatory drugs
* Recent serious bacterial, viral, fungal, or other opportunistic infections
* History of malignancy or serious uncontrolled cardiovascular, nervous system, pulmonary, renal, or gastrointestinal disease
* Serologic evidence of current or past viral infection: human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C, and human T-lymphotropic virus (HTLV) 1/2
* Positive QuantiFERON® tuberculosis (TB) test, purified protein derivative (PPD) skin test, history of tuberculosis, or active TB infection
* Active infection with Epstein-Barr Virus or Cytomegalovirus
* Liver disease
* Pregnant or breast-feeding
* Vaccination with a live virus within 8 weeks of receipt of study drug
* Vaccination with a killed virus within 2 weeks of receipt of study drug
* Participation in an investigational drug study within 90 days prior to screening
* Previously treated with a T-Reg based cell therapy
* History of allergy to gentamicin

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Losordo, MD, Study Director — Caladrius Biosciences
Locations (15):
- United States (15):
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Diabetes Research Institute, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Sanford Research, Fargo, North Dakota
  - Oregon Health Science University, Portland, Oregon
  - Sanford Research, Sioux Falls, South Dakota
  - Vanderbilt Eskind Diabetes Clinic, Nashville, Tennessee
  - Baylor College of Medicine / Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bender C, Wiedeman AE, Hu A, Ylescupidez A, Sietsema WK, Herold KC, Griffin KJ, Gitelman SE, Long SA; T-Rex Study Groupdagger; T-Rex Clinical Study Group. A phase 2 randomized trial with autologous polyclonal expanded regulatory T cells in children with new-onset type 1 diabetes. Sci Transl Med. 2024 May 8;16(746):eadn2404. doi: 10.1126/scitranslmed.adn2404. Epub 2024 May 8. PMID 38718135

RESULTS

PARTICIPANT FLOW:
Groups:
- CLBS03 Low Dose: A single infusion of CLBS03 Low Dose, a cell product comprised of autologous, ex vivo expanded regulatory T-cells resuspended in sterile USP (United States Pharmacopoeia) infusion solution.
  CLBS03 Low Dose
- CLBS03 High Dose: A single infusion of CLBS03 High Dose, a cell product comprised of autologous, ex vivo expanded regulatory T-cells resuspended in sterile USP infusion solution.
  CLBS03 High Dose
- Placebo: A single infusion of placebo, consisting of the infusion solution only
  Placebo
Period: Overall Study
Arm/Group | CLBS03 Low Dose | CLBS03 High Dose | Placebo
Started | 40 | 24 | 46
Completed | 37 | 22 | 43
Not Completed | 3 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLBS03 Low Dose | CLBS03 High Dose | Placebo | Total
Number analyzed (Participants) | 40 | 24 | 46 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 24 | 46 | 110
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 13 | 28
  Male | 30 | 19 | 33 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 2 | 9
  Not Hispanic or Latino | 34 | 22 | 44 | 100
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 3 | 5
  Black or African American | 1 | 0 | 1 | 2
  White | 36 | 23 | 42 | 101
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 24 | 46 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 4-hour Mixed Meal Tolerance Test (MMTT)-Stimulated C-peptide Area Under the Curve (AUC) at Week 52
Description: The area-under-curve of sequential C-peptide concentrations (AUC-Cpep) during the mixed-meal tolerance test (MMTT) is the gold-standard method to assess residual beta-cell (ie, insulin) secretion in type 1 diabetes.
Time Frame: Week 52
Measure: Mean (Standard Deviation); unit: pmol*hr/mL
Arm/Group | CLBS03 Low Dose | CLBS03 High Dose | Placebo
Number analyzed (Participants) | 40 | 24 | 46
pmol*hr/mL | -0.2863 (0.25988) | -0.3895 (0.31425) | -0.2670 (0.25745)

2. Secondary Outcome: Change From Baseline in 4-hour Mixed Meal Tolerance Test (MMTT)-Stimulated C-peptide Area Under the Curve (AUC) at Week 104
Description: as for outcome 1
Time Frame: Week 104
Measure: Mean (Standard Deviation); unit: pmol*hr/mL
Arm/Group | CLBS03 Low Dose | CLBS03 High Dose | Placebo
Number analyzed (Participants) | 40 | 24 | 46
pmol*hr/mL | -0.4492 (0.33135) | -0.5224 (0.33903) | -0.4412 (0.28923)

3. Secondary Outcome: Change in Hemoglobin A1c (HbA1c)
Time Frame: Week 104
Measure: Mean (Standard Deviation); unit: HbA1c %
Arm/Group | CLBS03 Low Dose | CLBS03 High Dose | Placebo
Number analyzed (Participants) | 39 | 24 | 46
HbA1c % | 1.56 (1.660) | 1.05 (1.474) | 1.77 (2.162)

4. Secondary Outcome: Change From Baseline in Mean Daily Dose of Insulin
Time Frame: Week 104
Measure: Mean (Standard Deviation); unit: U/kg body weight
Arm/Group | CLBS03 Low Dose | CLBS03 High Dose | Placebo
Number analyzed (Participants) | 39 | 24 | 46
U/kg body weight | 0.3840 (0.39727) | 0.4619 (0.40220) | 0.2874 (0.33602)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | CLBS03 Low Dose | CLBS03 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/24 | 0/46
Serious Adverse Events (participants affected / at risk) | 4/40 | 2/24 | 3/46
Other Adverse Events (participants affected / at risk) | 38/40 | 24/24 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLBS03 Low Dose (N=40) | CLBS03 High Dose (N=24) | Placebo (N=46)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CLBS03 Low Dose (N=40) | CLBS03 High Dose (N=24) | Placebo (N=46)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2
Nausea (Gastrointestinal disorders) | 4 | 1 | 2
Vomiting (Gastrointestinal disorders) | 5 | 2 | 10
Influence like illness (General disorders) | 2 | 2 | 2
Pyrexia (General disorders) | 3 | 2 | 3
Seasonal allergy (Immune system disorders) | 3 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 3
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 5
Influenza (Infections and infestations) | 4 | 3 | 4
Nasopharyngitis (Infections and infestations) | 7 | 8 | 7
Pharyngitis streptococcal (Infections and infestations) | 4 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 12 | 13 | 18
Viral infection (Infections and infestations) | 3 | 1 | 3
Concussion (Injury, poisoning and procedural complications) | 2 | 1 | 3
Limb injury (Injury, poisoning and procedural complications) | 3 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Headache (Nervous system disorders) | 8 | 5 | 11
Migraine (Nervous system disorders) | 0 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 2 | 1
Somnolence (Nervous system disorders) | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 2 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT02691247/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT02691247/SAP_001.pdf